CLINICAL TRIAL: NCT00908102
Title: The Prevalence of Low Back Symptoms in a Finnish Forestry Company - Effectiveness of Primary Care Interventions for Non-acute Low Back Symptoms in Occupational Health. Two Separate Randomised Controlled Trials (RCT) of Various Levels.
Brief Title: Managing Non-acute Low Back Symptoms in Occupational Health: Two Trials
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Helsinki (Other)
Collaborators: University of Oulu (Other); Juho Vainio Foundation (Other); Finnish Cultural Foundation (Other); Yrjo Jahnsson Foundation (Other); Finnish Work Environment Fund (Other)
Responsible Party: Principal Investigator, Jarmo Rantonen, MD, University of Helsinki
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: A18/01
Record Dates: First submitted 2009-05-19; First posted 2009-05-25 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Low Back Pain, Recurrent; Low Back Pain
Keywords: low back pain; recurrent; subacute; secondary prevention; primary care; occupational health; back book; rehabilitation
MeSH Terms: conditions — Low Back Pain; Recurrence

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- BB (Active Comparator): Subjects received the back book booklet, which is an self-information booklet about managing low back symptoms.
  Included in the Mild and Mild vs. NC interventions.
  Interventions: Other: Mild; Other: Mild vs. NC
- BB+A (Experimental): Subjects received a back book booklet and also oral advice based on the back book by the occupational health professional (OH Nurse or OH Physician in mild or moderate intervention, respectively).
  Included in the Mild and Mild vs. NC interventions. Arm was also used as a control at the Moderate and Moderate vs. NC interventions.
  Interventions: Other: Moderate; Other: Mild; Other: Mild vs. NC; Other: Moderate vs. NC
- DBC (Experimental): A graded activity back school program was carried out in a physiotherapy out-patient clinic that consisted of one-hour session twice or three times per week, lasting for 12 weeks, supervised by a specially trained physiotherapist. Arm is included in the MOderate and Moderate vs. NC interventions.
  Interventions: Other: Moderate; Other: Moderate vs. NC
- PMU (Experimental): An intensive, multidisciplinary LBP rehabilitation program was carried out in a physical medicine out-patient unit at the local Central Hospital. The program included a 3-week pre-course of 1,5 hour session at 3 days per week, closely followed by a 3-week intensive rehabilitation course of 6.5 hours per day for 5 days per week. A personal graded activity training program was made for each subject and patients were later called for follow-up visit within 1 year of the initial course. Arm is included in the MOderate and Moderate vs. NC interventions.
  Interventions: Other: Moderate; Other: Moderate vs. NC
- NC (Placebo Comparator): Natural course of low back pain
  Interventions: Other: Mild vs. NC; Other: Moderate vs. NC

INTERVENTIONS:
Other: Moderate — A two level active intervention with a control group was executed for patients suffering from non-acute, moderate LBP in occupational health. Patients were selected by using a self-administered postal questionnaire.
  Arms: BB+A; DBC; PMU
Other: Mild — A one level intervention with long-term effectiveness and cost-effectiveness was executed for patients suffering from non-acute mild level LBP in occupational health. Patients were selected by using a self-administered postal questionnaire.
  Arms: BB; BB+A
Other: Mild vs. NC — A two level intervention with long-term effectiveness and cost-effectiveness was executed for patients suffering from non-acute mild level LBP in occupational health. Intervention arms were compared to NC - no intervention group.
  Arms: BB; BB+A; NC
Other: Moderate vs. NC — A three level intervention with two control groups was executed for patients suffering from non-acute, moderate LBP in occupational health. RCT intervention groups were compared to NC group - i.e. no intervention.
  Arms: BB+A; DBC; NC; PMU

SUMMARY:
The purpose of this study is:

* Epidemiological part: characteristics of low back pain patients from a forestry company in Finland. Data is collected from occupational health databases and self administered questionnaires.
* Intervention: To determine the effectiveness and cost-effectiveness of several different interventions in subacute low back pain (LBP) patients in occupational health (OH).

DETAILED DESCRIPTION:
Eligible subjects were divided into two randomised controlled trials with the name of "mild" or "moderate" low back pain trials (interventions) and also mild vs natural course (NC) and moderate vs. NC interventions.

Pain, disability and quality of life were collected up to 2 years by self-administered questionnaires and sickness absences were gathered from electronical records for at least 4 year's follow up time.

ELIGIBILITY:
Inclusion Criteria:

* age 18-56 years
* present employment at the company
* at least one criteria out the following qualified for the study:

  * nonspecific LBP with the duration of 2 weeks or more
  * radiating, present low back pain
  * recurrent LBP (2 or more episodes per year)
  * work absence because of LBP
* included subjects also responded having low back pain during preceding week prior to the questionnaire (VAS ≥ 10 mm, Visual Analogue Scale 0-100 mm)

According to pain level, patients were later divided into two separate RCT's, "mild": VAS 10mm - 34mm, "moderate": VAS 35mm or more.

Exclusion Criteria:

* retirement
* acute nerve root compression symptoms
* malignant tumor
* recent fracture
* severe osteoporosis
* other specific disease preventing participation in the follow-up

Ages: 18 Years to 56 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 505 (Actual)
Dates: Start 2001-09; Primary Completion 2008-09 (Actual); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Sickness absence days (Low back (LB) specific, other than LB, total) | 6, 12, 24, 36, 48 months
Low back pain (VAS) | 0, 3, 6, 12, 24 months
Disability (Roland Morris 18) | 0, 3, 6, 12, 24 months
Quality of Life (15-D) | 0, 3, 6, 12, 24 months

SECONDARY OUTCOMES:
Sickness absence periods | 6, 12, 24, 36, 48 months
Disability (Oswestry's index) | 3, 6, 12, 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Simo Taimela, MD, docent, Study Director — Evalua Finland Co.; Jaro Karppinen, MD,professor, Study Director — University of Oulu; Markku Hupli, MD, PhD, Study Director — South Karelian Central Hospital; Jarmo O Rantonen, MD, Principal Investigator — University of Helsinki; Antti Malmivaara, MD, PhD, Study Director — Finnish Institute for Health and Welfare; Satu Luoto, MD, Study Director — South Karelian Central Hospital
Locations (1):
- University of Helsinki, Helsinki, Finland

REFERENCES:
- [Derived] Rantonen J, Karppinen J, Vehtari A, Luoto S, Viikari-Juntura E, Hupli M, Malmivaara A, Taimela S. Effectiveness of three interventions for secondary prevention of low back pain in the occupational health setting - a randomised controlled trial with a natural course control. BMC Public Health. 2018 May 8;18(1):598. doi: 10.1186/s12889-018-5476-8. PMID 29739371
- [Derived] Rantonen J, Karppinen J, Vehtari A, Luoto S, Viikari-Juntura E, Hupli M, Malmivaara A, Taimela S. Cost-effectiveness of providing patients with information on managing mild low-back symptoms in an occupational health setting. BMC Public Health. 2016 Apr 12;16:316. doi: 10.1186/s12889-016-2974-4. PMID 27068751
- [Derived] Rantonen J, Vehtari A, Karppinen J, Luoto S, Viikari-Juntura E, Hupli M, Malmivaara A, Taimela S. Face-to-face information combined with a booklet versus a booklet alone for treatment of mild low-back pain: a randomized controlled trial. Scand J Work Environ Health. 2014 Mar;40(2):156-66. doi: 10.5271/sjweh.3398. Epub 2013 Nov 1. PMID 24185642
- [Derived] Rantonen J, Luoto S, Vehtari A, Hupli M, Karppinen J, Malmivaara A, Taimela S. The effectiveness of two active interventions compared to self-care advice in employees with non-acute low back symptoms: a randomised, controlled trial with a 4-year follow-up in the occupational health setting. Occup Environ Med. 2012 Jan;69(1):12-20. doi: 10.1136/oem.2009.054312. Epub 2011 May 20. PMID 21602539